CLINICAL TRIAL: NCT02017301
Title: Influence of Acute Decompensation on Body Composition Determined by Bioelectrical Impedance Vector Analysis
Brief Title: Vector Analysis of Body Composition in Hospitalized Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Investigador Oficial, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: GAS-800-12-13-1
Record Dates: First submitted 2012-12-06; First posted 2013-12-20 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Infection
Keywords: Liver Cirrhosis,Infection, Impedance, Body Composition
MeSH Terms: conditions — Infections; Liver Cirrhosis | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Nutritional assessment — Daily nutritional assessment with bioelectrical impedance vector analysis, phase angle and mid-arm muscle circumference

SUMMARY:
Patients with acute decompensation of cirrhosis, or acute on chronic liver failure often present with malnutrition, and due to the in-hospital stay, their nutritional intake can vary widely, with several periods of fasting, and sometimes insufficient nutritional support. Therefore patients are prone to develop malnutrition or, the already present malnutrition worsens its status.

Our aim is to evaluate the daily changes in nutritional status in patients with acute decompensation of cirrhosis and evaluate the changes in plasma and serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Patients with confirmed cirrhosis.
* Any etiology
* Hospitalized with acute decompensation of cirrhosis
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Amputation
* Incomplete data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of hospitalized cirrhotic patients
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Changes in nutritional status | Daily measurement up to 30 days
  Nutritional status will be measured with bioelectrical impedance analysis (Vector and phase angle)

SECONDARY OUTCOMES:
Evaluation of inflammatory cytokines | Samples will be collected at the baseline evaluation.
  ELISA's test

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Astrid Ruiz-Margáin, M.Sc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubiran, México, D.F, Mexico

IPD SHARING:
Plan to Share IPD: No